CLINICAL TRIAL: NCT04787614
Title: 2019 National Survey of Early Care and Education (NSECE) COVID-19 Follow-up Study
Brief Title: 2019 NSECE COVID-19 Follow-up
Status: Completed | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Child Trends (Other); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rupa Datta, Distinguished Senior Fellow, National Opinion Research Center
Other Study IDs: HHSP233201500048I-CF
Record Dates: First submitted 2021-01-28; First posted 2021-03-08 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Child Care
Keywords: Early care and education; COVID-19; Center-based providers; Home-based providers; Caregivers; Child care; Workforce; ECE
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Home-based providers: Individuals who provided paid care for children under the age of 13 in a residential setting as of 2019
  Interventions: Other: No intervention
- Center-based providers: Providers who cared to children ages 0 through 5 years of age (not yet in kindergarten) in a non-residential setting as of 2019
  Interventions: Other: No intervention
- Center-based workforce: Individuals employed in center-based child care programs working directly with children in classrooms as of 2019
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of the National Survey of Early Care and Education (NSECE) is to document the nation's current supply of early care and education (ECE) services. Because the COVID-19 pandemic is likely to have had an impact on the ECE supply, and because the availability of ECE services is critical to restoring the U.S. economy, updated data on the ECE supply will be crucial for policy-making and research. The purpose of the NSECE COVID-19 Follow-up Study is to describe the impact of the COVID-19 pandemic on the pre-pandemic ECE supply and the ECE workforce, including changes in supply or departures from and re-entries to the workforce. Data from the study can be used to estimate the impact of the pandemic on ECE supply and the financial health of ECE providers, as well as providers' experiences during and after the pandemic emergency. Through a two-wave design, the NSECE COVID-19 Follow-up Study data will trace providers' and workforce members' experiences from 2019, through the initial months of the pandemic (to be reported in the Wave 1 interview), and then to the one-year point since the onset of the pandemic (to be reported in the Wave 2 interview). This design is intended to capture the trajectories of providers and workforce members, for example through recovery back to full or modified participation in ECE supply, or long-term exits from ECE supply. Prospectively collecting these data allows inference about the types of providers and workforce members most likely to have exited or survived in ECE, as well as the programmatic supports received by those who remain in ECE at the time of the second interview.

DETAILED DESCRIPTION:
The 2019 NSECE COVID-19 Follow-up Study includes three surveys: 1) NSECE COVID-19 Follow-up Home-based Provider Survey; 2) NSECE COVID-19 Follow-up Center-based Provider Survey; and 3) NSECE COVID-19 Follow-up Center-based Workforce Survey. This study aims to collect data from programs and individuals that completed interviews in the 2019 NSECE, regardless of whether or not they are still providing ECE services at the time of the follow-up surveys, with some exceptions (see Eligibility subsection below). The resulting data will document the experiences of ECE providers during the COVID-19 pandemic.

The study has a two-wave design, with surveys to be fielded in Fall 2020/Winter 2021 and Spring 2021. Wave 1 of the study includes all providers that completed interviews in 2019. For home-based providers and center-based workforce respondents, Wave 1 of the study will collect data from the same individuals interviewed in 2019. For center-based providers, Wave 1 of the study will collect data from center directors interviewed in 2019 or, if they are unavailable, other individuals knowledgeable about the center's operations. Wave 1 of the study will collect data on whether providers were still providing ECE services in February 2020, that is, prior to the pandemic emergency. Providers or center-based workforce members that had permanently ceased ECE services prior to February 2020 would not be fielded for Wave 2. Any providers or center-based workforce members who were participating in ECE provision at the onset of the pandemic will be fielded for Wave 2, so that trajectories of ECE participation, including temporary closures as well as permanent exits, can be identified in the Wave 2 interview. We note that home-based provider survey respondents are both ECE providers as well as members of the ECE workforce.

NSECE COVID-19 Follow-up Home-based Provider Survey. The purpose of this survey is to understand home-based providers' practices and statuses since March 2020, as well as personal impact on providers. The respondents for this survey include home-based providers who participated in the 2019 NSECE and reported getting paid for their work looking after children. The COVID-19 follow-up survey will ask home-based providers questions related to: 1) Employment Calendar (including the current status of the respondent's home-based program, employment changes and gaps since February 2020, and wages received) ; 2) Experience of Pandemic Assistance Programs (which will gather information about applications for program assistance, assistance received, and sources of information the respondent used to learn about child care and other types of assistance available); 3) ECE Practices during Reference Period (such as exposure to COVID-19, special health practices, and staffing and enrollment changes since March 2020/date of last interview); 4) ECE Status during Focal Week (covering items about cost of care, comprehensive services, and characteristics of the children enrolled during the last week of October 2020/April 2021); and 5) Current Personal Information (consisting of questions related to the respondent's current financial health, physical and mental health, household composition, and future ECE plans).

NSECE COVID-19 Follow-up Center-based Provider Survey. The purpose of this survey is to understand center practices and statuses since March 2020. The respondents for this survey include center-based providers who participated in the 2019 NSECE. The questionnaire will collect information on five topics: 1) Care Status Calendar (including the current status of the center-based organization, number of closures and openings since February 2020, reasons for closing, and reasons or conditions for reopening); 2) Experience of Pandemic Assistance Programs (applications for program assistance, assistance received, and sources of information the respondent used to learn about providing child care during the COVID-19 pandemic); 3) ECE Practices during Reference Period (including exposure to COVID-19, special health practices, types of contact with children when closed); 4) ECE Status during Focal Week (including items about cost of care, comprehensive services, program expenditures, and characteristics of staff and enrolled children during the last week of October 2020/April 2021); and 5) Current Personal Information (questions about the respondent's future ECE plans for themselves and for the organization as a whole).

NSECE COVID-19 Follow-up Center-based workforce Survey. The purpose of this survey is to understand ECE professional experiences and personal impact on ECE workers since March 2020. Respondents for this survey will include center-based classroom staff who completed the 2019 Center-based workforce questionnaire. The survey will include five sections: 1) Calendar (confirming employment status with center-based organization from 2019 NSECE); 2) Experience of Pandemic Assistance Programs (incorporating questions about questions about the sources of information the respondent used to learn about providing child care during and any special situations they may have worked under the COVID-19 pandemic) ; 3) ECE Practices during Reference Period (including information about any program exposure to COVID-19, special health practices, types of contact with children when closed, and any professional development activities during the pandemic); 4) ECE Status during Focal Week (information on the groups of children the respondent works with, child care activities planned, job stress, and center-based organizational support during the last week of October 2020/April 2021) ; and 5) Current Personal Information (asks questions about respondent's current financial health, physical and mental health, household composition, and future ECE plans).

ELIGIBILITY:
Inclusion Criteria:

* Completion of 2019 NSECE questionnaire

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The NSECE COVID-19 follow-up study population has been identified through the 2019 NSECE study. Listed home-based providers, paid unlisted home-based, center-based providers, and center-based workforce that have completed participated in the 2019 NSECE study will be asked to complete a questionnaire for the follow-up study. No additional participants will be considered during this data collection.
Sampling Method: Non-Probability Sample
Enrollment: 23472 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Impact of the COVID-19 pandemic on pre-pandemic supply of center-based care | 2020-2021 academic year
  The center-based provider questionnaire collects information periods of closure since the start of the pandemic to the time of the interview, experience with pandemic programs, ECE practices during reference period, ECE status during focal week.

SECONDARY OUTCOMES:
Impact of the COVID-19 pandemic on pre-pandemic supply of paid home-based care | 2020-2021 academic year
  The home-based provider questionnaire collects information on the provider's employment calendar, including periods of closure, experience with pandemic programs, ECE practices during reference period, ECE status during focal week, and current personal situation.

OTHER OUTCOMES:
Impact of the COVID-19 pandemic on pre-pandemic center-based provider workforce | 2020-2021 academic year
  The workforce questionnaire collects information about The workforce member's employment calendar, ECE practices during reference period, ECE status during focal week, and current personal situation.

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Datta, PhD, Principal Investigator — National Opinion Research Center
Locations (1):
- NORC at the University of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: National Survey of Early Care and Education 2019: 2017 - 2022 - Overview — https://www.acf.hhs.gov/opre/project/national-survey-early-care-and-education-2019-2017-2022-overview